CLINICAL TRIAL: NCT05467631
Title: Topical Phytoterpene Mixture for Treatment of Plantar Fasciitis in Adults
Brief Title: Topical Phytoterpenes for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Biomedical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PF-001
Record Dates: First submitted 2021-10-26; First posted 2022-07-20 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Plantar Fasciitis
Keywords: Heel pain; plantar; fasciitis; foot pain
MeSH Terms: conditions — Fasciitis, Plantar; Fasciitis

STUDY DESIGN:
Intervention Model Description: 2 groups, plain tea tree oil control and formulated essential oil blend with permeation enhancer as treatment in a randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical bottles given to participants with serial number, aroma and feel of each treatment group is the same
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain Tea Tree Oil Control (Active Comparator): Topical application of 1ml 20% tea tree oil in almond oil base as a carrier twice daily for 2 weeks.
  Interventions: Other: Topical oil application
- Verum (Experimental): Topical application twice daily of 1ml mixture for 2 weeks of essential oils containing tea tree oil, rosemary, clove, pepper, in a formulation with skin permeation enhancers including limonene.
  Interventions: Other: Topical oil application

INTERVENTIONS:
Other: Topical oil application — Topical Comparison

SUMMARY:
Randomized controlled trial of mixture of essential oils containing tea tree oil, rosemary, clove, pepper, in a formulation with skin permeation enhancers including limonene for the treatment of plantar fasciitis in adult men and women. Forty-two patients will be randomized to receive twice daily topical application of the treatment formulation or plain tea tree oil as a control. Analog pain scores will be assessed at the start of treatment and at two weeks. Analysis will be by student's T-test.

DETAILED DESCRIPTION:
Randomized controlled trial of mixture of essential oils containing tea tree oil, rosemary, clove, pepper, in a formulation with skin permeation enhancers including limonene for the treatment of plantar fasciitis in adult men and women. Forty-two patients will be randomized to receive twice daily topical application of the treatment formulation or plain tea tree oil as a control. Analog pain scores will be assessed at the start of treatment and at two weeks. Analysis will be by student's T-test. Primary outcome measure will be the difference in pain score between baseline score and pain score at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Plantar fasciitis diagnosed by a medical practitioner and at least 3 months in duration

Exclusion Criteria:

* Age under 18 years, any history of diabetes, history of foot surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score Between Baseline and 2 Weeks | 2 weeks
  Patients will be asked to rate pain on a 1-10 analog scale at the start of the study and at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Briant Burke, MD, Principal Investigator — Center for Biomedical Research, Inc.
Locations (1):
- Center for Biomedical Research,Inc., Boise, Idaho, United States

REFERENCES:
- [Derived] Burke BE, Baillie JE. Randomized placebo controlled trial of phytoterpenes in DMSO for the treatment of plantar fasciitis. Sci Rep. 2024 Jul 31;14(1):17621. doi: 10.1038/s41598-024-65979-1. PMID 39085322